CLINICAL TRIAL: NCT02111109
Title: An Observational Pilot Study of the Effects of Traumatic Haemorrhagic Shock and Resuscitation on the Microcirculation
Acronym: MICROSHOCK
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 14/YH/0078
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Traumatic Haemorrhagic Shock
Keywords: Microcirculation; Trauma; Haemorrhage; Shock
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood / plasma / urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Traumatic injury
  Interventions: Device: Side Stream Dark Field Microscopy

INTERVENTIONS:
Device: Side Stream Dark Field Microscopy

SUMMARY:
Haemorrhage following major trauma is an important preventable cause of death. Those patients who survive may have a prolonged period of debility caused by failure of key body organs. We suspect that an important contributor to this organ failure may be dysfunction in the network of small blood vessels that supply the bodies organs with oxygen and nutrients. Our study will examine the link between the microcirculation and organ failure in patients who have suffered significant bleeding after traumatic injury. We will also explore the relationship between resuscitation of the global circulation (blood pressure, cardiac output etc.)an area that is monitored in clinical practice with the state of the microcirculation, which by contrast is not monitored. Patients with severe traumatic injury commonly have problems with blood clotting. Some researchers have suggested that microcirculatory failure may be an important contributor to this problem and we will explore this in more detail. Finally, we will attempt to examine some of the mechanisms by which the microcirculation may be disrupted by trauma and subsequent bleeding. These may include inappropriate activation of white blood cells, inadequate function of oxygen carrying red blood cells and changes to the cells lining the small blood vessels.

We will use a non invasive method to assess the microcirculation termed Side Stream Dark Field microscopy. This involves recorded a video image of the movement of blood within the small blood vessels under a patients tongue. In addition we will use ultrasound to assess the flow of blood from the heart. Small samples of blood will be taken to assess blood clotting and to look at possible mechanisms of microcirculatory dysfunction.

We aim to study ten patients in the first instance. The study will be carried out within the intensive care units at Kings College Hospital.

ELIGIBILITY:
Inclusion Criteria History of traumatic injury received blood products prior to ICU admission

Exclusion Criteria:

Not expected to survive 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with traumatci injury, haemorrhae and impaired perfusion
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2014-07; Primary Completion 2017-05 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
SOFA score | 72 hours

SECONDARY OUTCOMES:
Length of ICU stay | 28 days
Mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - University Hospital Birmingham, Birmingham, West Midlands
  - Kings College Hospital, London
  - Royal London Hospital, London

REFERENCES:
- [Derived] Naumann DN, Hazeldine J, Midwinter MJ, Hutchings SD, Harrison P. Poor microcirculatory flow dynamics are associated with endothelial cell damage and glycocalyx shedding after traumatic hemorrhagic shock. J Trauma Acute Care Surg. 2018 Jan;84(1):81-88. doi: 10.1097/TA.0000000000001695. PMID 28885470
- [Derived] Naumann DN, Mellis C, Smith IM, Mamuza J, Skene I, Harris T, Midwinter MJ, Hutchings SD. Safety and feasibility of sublingual microcirculation assessment in the emergency department for civilian and military patients with traumatic haemorrhagic shock: a prospective cohort study. BMJ Open. 2016 Dec 21;6(12):e014162. doi: 10.1136/bmjopen-2016-014162. PMID 28003301
- [Derived] Hutchings S, Naumann DN, Harris T, Wendon J, Midwinter MJ. Observational study of the effects of traumatic injury, haemorrhagic shock and resuscitation on the microcirculation: a protocol for the MICROSHOCK study. BMJ Open. 2016 Mar 4;6(3):e010893. doi: 10.1136/bmjopen-2015-010893. PMID 26944694